CLINICAL TRIAL: NCT02216084
Title: BAX930 (rADAMTS13): A Phase 1 Prospective, Uncontrolled, Open-Label, Multicenter, Dose-Escalation Study Evaluating the Safety and Pharmacokinetics in Hereditary Thrombotic Thrombocytopenic Purpura (TTP)
Brief Title: Phase 1 Dose Escalation, Single Dose Study to Assess Safety and Pharmacokinetics of BAX930 in Hereditary Thrombotic Thrombocytopenic Purpura (TTP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 281101; 2012-003221-19 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Thrombotic Thrombocytopenic Purpura (TTP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant ADAMTS13 (Experimental): The study is comprised of 3 dose cohorts and two dose escalation steps [Cohort 1: 3 subjects; Cohort 2: 3 subjects; Cohort 3: 8 subjects]. Subjects will be enrolled and dosed sequentially. Subjects will be recruited to the next dose level only after short-term safety has been demonstrated and reviewed by an independent Data Monitoring Committee (DMC) at the preceding dose level. The first 2 subjects in any cohort will be ≥ 18 years of age. The effects of the investigational product on vital signs, hematology, and clinical chemistry parameters (up to 96 ± 2 hrs blood sampling timepoint) will determine short-term safety. The DMC will recommend whether to proceed with the study or in case of a safety concern recommend remedial actions and/or to discontinue the study. Subject participation will continue until 28 ± 3 days after infusion of the investigational product. Subject participation in one Dose Cohort (1-3) is expected to be approximately 6-8 weeks.
  Interventions: Drug: Recombinant ADAMTS13

INTERVENTIONS:
Drug: Recombinant ADAMTS13 — rADAMTS13 (a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13) is a lyophilized formulation for intravenous injection. The lyophilized rADAMTS13 is reconstituted with sterile water for injection.
  Subjects will receive an intravenous injection with rADAMTS13 at a dose of either 5 U/kg bodyweight (Cohort 1), or 20 U/kg bodyweight (Cohort 2), or 40 U/kg bodyweight (Cohort 3).

SUMMARY:
The purpose of this Phase 1, prospective, uncontrolled, open-label, multicenter, dose-escalation study is to evaluate the safety, including immunogenicity, and pharmacokinetics of BAX930 (rADAMTS13) in a total of 14 evaluable subjects diagnosed with severe hereditary thrombotic thrombocytopenic purpura (TTP) (plasma ADAMTS13 activity <6%) who are assigned to one of three dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 12 and 65 years of age, inclusive. (The first 2 subjects in any cohort will be ≥ 18 years of age.)
* Subject and/or legally authorized representative has provided written informed consent.
* Subject has a documented diagnosis of severe hereditary ADAMTS13 deficiency, defined as 1) confirmed by genetic testing, documented in patient history or at screening, and 2) ADAMTS13 activity < 6%, documented in patient history or at screening. NOTE: In patients receiving prophylactic therapy with fresh frozen plasma (FFP) or other ADAMTS13 containing products, the levels of plasma ADAMTS13 activity may exceed 6% at screening.
* Cryoprecipitate, FFP, or other ADAMTS13 containing products interfering with ADAMTS13 PK have to be paused at least 10 days prior to infusion of the investigational product.
* The subject is not displaying any severe TTP symptoms at screening. Patients presenting with minor, but stable laboratory abnormalities (LDH not higher than 3 times the upper limit of normal; platelet count not lower than 100,000 per μl) at screening may be enrolled.
* Subjects ≥18 years of age have a Karnofsky score ≥ 60%, and subjects < 18 years of age have a Lansky score ≥ 70%.
* Subject is hepatitis C virus negative (HCV-) as confirmed by antibody or polymerase chain reaction (PCR) testing; HCV positive (HCV+) subjects are eligible for inclusion if their disease is chronic but stable.
* If female of childbearing potential, subject presents with a negative serum pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
* Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Subject has been diagnosed with any other TTP-like disorder (for example, microangiopathic hemolytic anemia), including acquired TTP.
* Subject has known hypersensitivity to hamster proteins or other components of the investigational product.
* Subject has a medical history or presence of a functional neutralizing ADAMTS13 inhibitor at screening.
* Subject has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis/mild asthma, food allergies or animal allergies.
* Subject has a medical history of hematological disorders, in particular systemic lupus erythematosus, amyloidosis, antiphospholipid antibody syndrome, vasculitis, other hemolytic anemia, disseminated intravascular coagulation, and systemic scleroderma.
* Subject has a history of significant neurological events, such as major stroke, indicating that a relapse might have severe consequences, as judged by the investigator.
* Subject is HIV positive with an absolute CD4 count < 200/mm3.
* Subject has been diagnosed with a cardiovascular disease [New York Heart Association (NYHA) classes 3-4].
* Subject is scheduled to undergo elective surgery during study participation.
* Subject has been diagnosed with severe liver disease, as evidenced by, but not limited to, any of the following: serum ALT 3 times the upper limit of normal, international normalized ratio (INR) > 1.5, hypoalbuminemia, portal vein hypertension (e.g. presence of otherwise unexplained splenomegaly, history of esophageal varices).
* Subject has been diagnosed with severe glomerular disease, with gross proteinuria and a serum creatinine level ≥ 2.5 mg/dL.
* Subject has been treated with an immunomodulatory drug, in case of corticoids with an equivalent to hydrocortisone greater than 10 mg /day, excluding topical treatment (e.g. ointments, nasal spray), within 30 days prior to enrollment.
* Subject has a history of drug and/or alcohol abuse within the last 6 months prior to study enrollment.
* Subject has a life expectancy of less than 3 months.
* Subject is identified by the investigator as being unable or unwilling to cooperate with study procedures.
* Subject is a family member or employee of the investigator.
* Subject suffers from a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
* If female, subject is pregnant or lactating at the time of study enrollment.
* Subject has participated in another clinical study involving an investigational product or device within 30 days prior to study enrollment.
* Subject is scheduled to participate in another clinical study involving an investigational product or device during the course of this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (serious and non-serious), including the incidence of binding and inhibitory antibody formation | Up to 28 (± 3) days after investigational product infusion

SECONDARY OUTCOMES:
Pharmacokinetic [PK] parameter 'incremental recovery [IR]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'maximum concentration following infusion [Cmax]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'minimum time to reach Cmax [T max]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'terminal or disposition half-life [T1/2]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'mean residence time [MRT]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'systemic clearance [Cl]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'area under the plasma/time curve [AUC]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
PK parameter 'steady state volume of distribution [Vss]' | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3
Plasma von Willebrand factor: Ristocetin cofactor activity [VWF:RCo], von Willebrand factor antigen [VWF:Ag] and VWF structure analysis | Within 1 hour pre-infusion and up to 288 (± 4) hours post-infusion
  Will be evaluated after single infusions of rADAMTS13 in Dose Cohorts 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (3):
  - Ohio State University Medical Center, Dublin, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Methodist Hospital Research Institute, Houston, Texas
- General Hospital Vienna (Allgemeines Krankenhaus der Stadt Wien), Vienna, Austria
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
- Japan (2):
  - • Tokyo Medical and Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Hyogo College of Medicine Hospital, Department of Hematology, Nishinomiya-shi
- Institute of Hematology and Transfusion Medicine, Warsaw, Poland
- Inselspital - Universitaetsspital Bern, Bern, Switzerland
- University College London Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Scully M, Knobl P, Kentouche K, Rice L, Windyga J, Schneppenheim R, Kremer Hovinga JA, Kajiwara M, Fujimura Y, Maggiore C, Doralt J, Hibbard C, Martell L, Ewenstein B. Recombinant ADAMTS-13: first-in-human pharmacokinetics and safety in congenital thrombotic thrombocytopenic purpura. Blood. 2017 Nov 9;130(19):2055-2063. doi: 10.1182/blood-2017-06-788026. Epub 2017 Sep 14. PMID 28912376